CLINICAL TRIAL: NCT01605370
Title: Can Nebivolol Reverse Inappropriate Left Ventricular Mass in Hypertensive Patients?
Acronym: Inapprop
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in identifying subjects satisfying the inclusion criteria.
Sponsor: Mayo Clinic (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Marek Belohlavek, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-007035
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Hypertension
Keywords: Hypertension, Left Ventricular Mass
MeSH Terms: conditions — Hypertension | interventions — Nebivolol; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebivolol (Experimental): Subjects randomized to this arm will receive Nebivolol 2.5 mg once daily.
  Interventions: Drug: Nebivolol
- Metoprolol succinate (Other): Subjects randomized to this arm will receive metoprolol succinate 50 mg once daily.
  Interventions: Drug: Metoprolol succinate

INTERVENTIONS:
Drug: Nebivolol — Nebivolol 2.5 mg once daily
  Other Names: Bystolic
  Arms: Nebivolol
Drug: Metoprolol succinate — Metoprolol succinate 50 mg once daily
  Other Names: Toprol XL
  Arms: Metoprolol succinate

SUMMARY:
The purpose of this study is to evaluate if a drug called nebivolol can reverse inappropriate left ventricular mass (LVM) when compared to the standard of care drug metoprolol.

DETAILED DESCRIPTION:
In response to chronic pressure overload by arterial hypertension, the cardiac left ventricle undergoes hypertrophy, that is, increases its wall thickness and, therefore, its mass, to sustain the elevated workload. Such anatomical remodeling can be considered adaptive or appropriate. However, in a considerable number of patients with arterial hypertension, the increase in the left ventricular mass is excessive and, thus, inappropriate.

Ventricular mass is inappropriate when its amount surpasses the physical need of the ventricle to sustain the elevated workload. Therefore, ventricular mass can be inappropriate even in patients without arterial hypertension or without hypertrophy identified by echocardiography (echo). We can mathematically predict an appropriate amount of mass and observe the actual mass in individual patients based on ventricular workload and wall thickness, respectively, noninvasively evaluated by echo. By comparing the observed ventricular mass to the predicted one, we determine whether its amount is inappropriate. It follows that by therapeutically normalizing blood pressure in hypertension and thus eliminating the elevated workload, then any ventricular hypertrophy represents an inappropriate mass.

Inappropriate ventricular mass is proven to have a detrimental effect on long-term cardiovascular event-free survival, and ventricular hypertrophy is increasingly recognized as a potent risk factor of cardiovascular morbidity and mortality, and all-cause mortality. Ventricular performance is altered in hypertension with inappropriate mass, but this alteration can be subtle enough to escape detection using current echocardiography measures. Hence, patients with hypertension, who have inappropriate left ventricular mass, need to be specifically identified by analysis of the predicted and observed ventricular mass, and the therapeutic goal must include management of elevated blood pressure as well as reversal of the excessive ventricular mass.

In this double-blind prospective study, patients with hypertension and inappropriate ventricular mass will be randomized to therapy with nebivolol or metoprolol to find out whether nebivolol could reverse inappropriate left ventricular mass, thus providing a benefit beyond what is achieved by mere blood pressure reduction alone. If confirmed, this will represent a significant ancillary ability of nebivolol and be a key step towards therapy of inappropriate ventricular mass, which is a so far unmanaged cardiovascular risk and a poor event-free prognostic factor.

ELIGIBILITY:
All candidates must have previously untreated hypertension. The candidates will be picked from patients with stage-1 hypertension (systolic BP 140-159 mm Hg or diastolic BP 90-99 mm Hg) and those with stage-2 hypertension (systolic BP ≥160 mm Hg or diastolic BP ≥100), based on the seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure guidelines (JNC-7).

Inclusion Criteria:

* Presence of inappropriate LVM.
* Presence of phenotype of inappropriate LVM.

Exclusion Criteria:

The criteria will assure that only patients with hypertension are enrolled, that is, excluded will be subjects with systolic BP < 140 or diastolic BP < 90 (ie, prehypertension or normal BP), but without complications or any indication (or suspicion) of end-organ damage based on a physical exam, clinical history, or laboratory tests.

Specific exclusion criteria are:

* Reactive airways disease including asthma.
* Diabetes mellitus or hypoglycemia; thyrotoxicosis.
* LV dysfunction (ejection fraction < 50%) or heart failure.
* Present or previously documented coronary heart disease or angina.
* Acute myocardial infarction, or history of myocardial infarction.
* Severe bradycardia, heart block greater than first degree or sick sinus syndrome (unless a permanent pacemaker is in place).
* Hepatic insufficiency or history of cirrhosis.
* Chronic renal failure or renovascular dysfunction.
* Cerebrovascular dysfunction.
* Peripheral vascular disease.
* Pregnant or nursing women; women of childbearing age will be required to take a pregnancy test at the time of enrollment and use an acceptable method of birth control.
* Poor echo image quality.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marek Belohlavek, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Scottsdale, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nebivolol | Metoprolol Succinate
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated early due to the difficulty in identifying subjects satisfying the inclusion criteria. Only 1 subject was enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Metoprolol Succinate | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Gender [Number; unit: participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Inappropriate Left Ventricular Mass (LVM)
Description: LVM will be measured by echocardiography exam. LVM is inappropriate when observed LVM (oLVM) exceeds predicted LVM (pLVM) by more than 28%, that is, 100×(oLVM/pLVM) >128%.
Time Frame: baseline, 6 months
Population: Data were not collected for the single participant, so no analysis was performed.
Arm/Group | Nebivolol | Metoprolol Succinate
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Nebivolol | Metoprolol Succinate
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nebivolol (N=1) | Metoprolol Succinate (N=0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early due to the difficulty in identifying subjects satisfying the inclusion criteria. Only 1 subject was enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No